CLINICAL TRIAL: NCT01806948
Title: Efficacy Study of Antiemetics to Reduce Postoperative Nausea and Vomiting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kidong Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SNUBH_GO_017
Record Dates: First submitted 2013-03-06; First posted 2013-03-07 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — ramosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Single dose of antiemetics. Specifically, Ramosetron 0.3 mg will be intravenously injected when surgery is ended. Additionally, placebo will be intravenously injected at 4 hours after surgery.
  Interventions: Drug: Ramosetron
- Experimental (Experimental): Double dose of antiemetics. Specifically, Ramosetron 0.3 mg will be intravenously injected when surgery is ended. Additionally, Ramosetron 0.3 mg will be intravenously injected at 4 hours after surgery.
  Interventions: Drug: Ramosetron

INTERVENTIONS:
Drug: Ramosetron

SUMMARY:
We randomized patients who received laparoscopic surgery for benign gynecologic disease into double dose (Experimental Group) or single dose (Control Group) of antiemetics. We compared the degree of postoperative nausea and vomiting in experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopy for benign gynecologic disease

Exclusion Criteria:

* Vomiting within 24 hours before surgery
* Not using patient controlled analgesics postoperatively

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Complete Response Rate | Postoperative 24 hours
  The percentage of patients who experienced neither nausea nor vomiting within 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea